CLINICAL TRIAL: NCT05272345
Title: Follow-Up Wıth Dıagnosıs Of Fıbromyalgıa In Patıents Wıth Sexual Functıonal Dısorder Evaluatıon Of Sexual Therapy And Post-Therapy Fıbromyalgıa
Brief Title: Fibromyalgia and Sexual Functıonal Dısorder and Sexual Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Pinar Kadiroğulları Principal investigator , DEPARTMENT OF OBSTETRICS AND GYNECOLOGY, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK/2022-03
Record Dates: First submitted 2022-02-13; First posted 2022-03-09 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Fibromyalgia; Sexual Dysfunction
Keywords: Fibromyalgia; Patients; Quality of Life; Sexual desire; FSFI scala
MeSH Terms: conditions — Fibromyalgia; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fibromyalgia status before sexual therapy/ Fibromyalgia condition after sex therapy (Experimental): * Women with sexual dysfunction (FSFI score < 26.55) in reproductive age (15-49 years) followed up with a diagnosis of fibromyalgia
  * Women with sexual dysfunction (FSFI score < 26.55) in reproductive age (15-49 years) followed up with a diagnosis of fibromyalgia and who were reevaluated for fibromyalgia after sexual therapy was given
  Interventions: Procedure: sexual therapy

INTERVENTIONS:
Procedure: sexual therapy — In sexual therapy; A total of 4 sessions of therapy were initiated with the patients, one session per week for 1 month.

SUMMARY:
investigators aim to re-evaluate the findings of Fibromyalgia in patients whose FSFI scores return to normal levels after sexual therapy, by identifying patients with sexual dysfunction according to the FSFI scale applied in patients investigators followed up with a diagnosis of fibromyalgia, and when investigators consulted with obstetricians.

DETAILED DESCRIPTION:
Apart from routine Fibromyalgia treatments, investigators think that Fibromyalgia patients should be evaluated in detail in terms of sexual dysfunction, and better results will be obtained by adding sexual therapy to the treatment in patients with FSFI score below 26.55.

In the current literature review, investigators have seen that there is no study on the evaluation of fibromyalgia before and after sexual therapy.

investigators think that our study will be a pioneer in terms of showing the importance of the multidisciplinary approach in the treatment of Fibromyalgia.

investigators foresee that sexuality is still a subject that is avoided to be talked about due to the cultural infrastructure of developing countries, and that Fibromyalgia will actually decrease with the regulation of sexual life.

investigators believe that more comprehensive studies with this perspective will develop a multidisciplinary approach in Fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Follow-up with a diagnosis of fibromyalgia
* Reproductive age (15-49 years)
* Women with sexual dysfunction (FSFI score < 26.55)

Exclusion Criteria:

* Women Wıth Ibromyalgıa Wıthout Sexual Dysfunction
* Women Wıth A Score Greater 26.55 Wıthout Therapy

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2025-12-14 (Estimated)

PRIMARY OUTCOMES:
VAS evaluation results for pain before sexual therapy in patients with fibromyalgia | 6 months
  Evaluation results of women with fibromyalgia diagnosis with VAS SCAL VAS SCALE; THE PATIENT IS REQUESTED TO VALUE THE PAIN BETWEEN 0-10. 0 ; NO PAIN 10: SEVERE PAIN
VAS evaluation results for pain after sexual therapy in patients with fibromyalgia | 6 months
  Evaluation results of women with fibromyalgia diagnosis with VAS SCAL after sexual therapy VAS SCALE; THE PATIENT IS REQUESTED TO VALUE THE PAIN BETWEEN 0-10. 0 ; NO PAIN 10: SEVERE PAIN
FSFI scores before sexual therapy in patients with fibromyalgia | 6 months
  Evaluation results of women with fibromyalgia diagnosis with FSFI SCAL
  * The FSFI questionnaire consists of 19 questions; It evaluates 6 main factors as sexual desire, sexual arousal, lubrication, orgasm, satisfaction and pain/discomfort. The highest total raw score that can be obtained in this scale is 95, the lowest raw score is 4, and the highest score is 36 after the product of the coefficients, and the lowest score is 2. Effect coefficients used for scoring the whole scale; 0.6 for sexual desire, 0.3 for sexual arousal and lubrication, and 0.4 for orgasm, satisfaction, and pain/discomfort. A FSFI score below 26.55 was defined as compatible with sexual dysfunction.
FSFI scores after sexual therapy in patients with fibromyalgia | 6 months
  Evaluation results of women with fibromyalgia diagnosis with FSFI SCAL after sexual therapy
  * The FSFI questionnaire consists of 19 questions; It evaluates 6 main factors as sexual desire, sexual arousal, lubrication, orgasm, satisfaction and pain/discomfort. The highest total raw score that can be obtained in this scale is 95, the lowest raw score is 4, and the highest score is 36 after the product of the coefficients, and the lowest score is 2. Effect coefficients used for scoring the whole scale; 0.6 for sexual desire, 0.3 for sexual arousal and lubrication, and 0.4 for orgasm, satisfaction, and pain/discomfort. A FSFI score below 26.55 was defined as compatible with sexual dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Kadiroğulları, Principal Investigator — Acıbadem University Atakent Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Acıbadem University Atakent Hospital, Department of Obstetrics and Gynecology,, Istanbul
  - Pınar Kadiroğulları, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided